CLINICAL TRIAL: NCT02156063
Title: A Randomised, Double Blind, Multi-center, Placebo-controlled Study to Evaluate the Efficacy, Safety, and Tolerability of NT100 in Pregnant Women With a History of Unexplained Recurrent Pregnancy Loss (RPL)
Brief Title: A Multi-center, Placebo-controlled Study to Evaluate NT100 in Pregnant Women With a History of Unexplained Recurrent Pregnancy Loss (RPL)
Acronym: RESPONSE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nora Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NT-05
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Recurrent Pregnancy Loss; Recurrent Miscarriage
Keywords: Recurrent Pregnancy Loss; Recurrent Miscarriage; Miscarriage; Pregnancy Loss; Repeated Pregnancy Loss
MeSH Terms: conditions — Abortion, Habitual; Abortion, Spontaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NT100 (Experimental): NT100 Dose 1
  Interventions: Drug: NT100
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NT100
  Arms: NT100
Drug: Placebo
  Arms: Placebo

SUMMARY:
This is a randomised, double blind, multi-center, placebo-controlled study of subcutaneous NT100 in pregnant women with a history of unexplained recurrent pregnancy loss. Approximately 150 participants will be randomised to receive subcutaneous NT100 or placebo.

DETAILED DESCRIPTION:
This is a randomised, double blind, multi-center, placebo-controlled study of subcutaneous NT100 in pregnant women with a history of unexplained recurrent pregnancy loss. Approximately 150 participants will be randomised to receive subcutaneous NT100 or placebo. Participants will be screened for eligibility, and will begin attempts at spontaneous conception. Following randomization and initiation of study drug treatment, participants will visit the study site at specified intervals throughout the study for assessments and blood work.

All participants will be monitored for adverse events. All participants who have received at least one dose of study drug will be followed for safety for a minimum of 4 weeks following the last dose of study drug. After delivery, pregnancy outcome information will be obtained.

ELIGIBILITY:
Inclusion Criteria:

1. Pre-menopausal female 18-37 years of age at consent, trying to conceive
2. Documented history of unexplained recurrent pregnancy loss
3. Spontaneous conception, as confirmed by urine pregnancy test performed at the investigative site
4. Body mass index (BMI) of 19-35 kg/m2 at consent

Exclusion Criteria:

1. Greater than 5 weeks of gestation when presenting for randomisation.
2. Known karyotype abnormalities in either the participant or her current male partner
3. Uncorrected clinically significant intrauterine abnormalities
4. Abnormal vaginal bleeding of unknown cause
5. Current diagnosis of infertility in either the participant or her current male partner
6. Current or past diagnosis of systemic autoimmune disease, coagulopathy, hyperprolactinemia, cervical incompetence, or high-grade cervical dysplasia with conization/surgery.
7. Any uncontrolled clinically significant medical condition

Ages: 18 Years to 37 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-06; Primary Completion 2016-01 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Pregnancy | at Week 20 of gestation
  The primary outcome measure is clinical pregnancy at Week 20 of gestation

SECONDARY OUTCOMES:
Live birth | at any time during pregnancy
Clinical pregnancy | at Weeks 6, 8 and 12 of gestation
Spontaneous pregnancy loss | within 24 weeks of gestation
Stillbirth | after 24 weeks of gestation
Subjects with adverse events and serious adverse events | during treatment and within 4 weeks after treatment
Changes in clinical laboratory parameters following study drug exposure | during treatment and within 4 weeks after treatment

CONTACTS AND LOCATIONS:
Locations (19):
- United Kingdom (19):
  - Ashington
  - Birmingham
  - Chertsey, Surrey
  - Coventry
  - Edinburgh
  - Frimley, Surrey
  - Leeds
  - Liverpool
  - London
  - Manchester
  - Middlesbrough
  - Newcastle upon Tyne
  - Nottingham
  - Oxford
  - Plymouth
  - South Shields
  - Southamptom
  - Stoke-on-Trent
  - Sunderland

REFERENCES:
- [Derived] Eapen A, Joing M, Kwon P, Tong J, Maneta E, De Santo C, Mussai F, Lissauer D, Carter D; RESPONSE study group. Recombinant human granulocyte- colony stimulating factor in women with unexplained recurrent pregnancy losses: a randomized clinical trial. Hum Reprod. 2019 Mar 1;34(3):424-432. doi: 10.1093/humrep/dey393. PMID 30776296